CLINICAL TRIAL: NCT04691245
Title: Three Dimensional Ultrasound Guided Femoral Access for Transcatheter Aortic Valve Implantation
Brief Title: 3D US Guided Femoral Artery Access for TAVI
Acronym: 3D-US-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Harm Scholten, md, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3D-US-TAVI
Record Dates: First submitted 2020-12-20; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Ultrasound Therapy; Complications; Femoral Artery Injury
Keywords: 3D Ultrasound; vascular access; Transcatheter aortic valve implantation

STUDY DESIGN:
Intervention Model Description: randomized clinical trial with two arms
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Femoral access using 3D US
  Interventions: Device: 3D US
- Control (Active Comparator): Femoral access using 2D US
  Interventions: Device: 2D US

INTERVENTIONS:
Device: 3D US — 3D US guided access to femoral artery
  Arms: Intervention
Device: 2D US — 2D US guided access to femoral artery
  Arms: Control

SUMMARY:
Rationale: Bleeding and vascular complications of the femoral artery still account for significant morbidity and mortality in transcatheter aortic valve implantation procedures. Although steadily declining over the past years through smaller diameter devices and use of ultrasound, major complications still occur in 3-4 % of patients. Femoral access is often obtained using 2D US guidance already. New 3D US probes can aid in increasing anatomical awareness. This can improve first pass success during procedures. Furthermore, for new closure devices, entering the artery at a straight angle at precisely 12 o'clock probably reduces complications. Therefore, the investigators hypothesize improved real time needle guidance using three dimensional ultrasound can decrease procedure related complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult age (>18 years)
* Scheduled to undergo elective transcatheter aortic valve implantation with percutaneous access through the femoral artery
* Written Informed consent

Exclusion Criteria:

* Unable to obtain informed consent
* Vascular access via alternative approach (radial/subclavian) or surgical cutdown

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
first pass success | during procedure/surgery
  successful entry in femoral artery within one skinbreak and without needle redirections

SECONDARY OUTCOMES:
imaging time | during procedure/surgery
  time from putting probe on skin to start procedure (in seconds)
procedure time | during procedure/surgery
  time from puncturing skin until entry in femoral artery (in seconds)
total number of punctures | during procedure/surgery
  new skin breaks needed for completion of procedure
number of needle redirections | during procedure/surgery
  total number of needle withdrawals >5mm but without needing new skin puncture
12 o clock entry | during procedure/surgery
  entrance to femoral artery at exactly 12 o clock (antero-medial)
needle visualization | during procedure/surgery
  rated from good-adequate-poor
operator satisfaction | during procedure/surgery
  likert scale 1-5 with 1 no satisfaction and 5 completely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No